CLINICAL TRIAL: NCT03838536
Title: Synergistic Activity of Choline, Lutein, and Docosahexaenoic Acid in Human Milk in Support of Cognitive Development: An Egg Intervention Feasibility Study
Brief Title: Synergistic Activity of Human Milk Nutrients and Infant Cognition
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Egg Nutrition Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 18-2216
Record Dates: First submitted 2019-02-05; First posted 2019-02-12 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Breastfeeding, Exclusive
Keywords: Breastfeeding; Eggs; Baby
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to whole egg or egg white powder to consume throughout the study.
Who Masked: Participant
Masking Description: The participants will be given a jar of egg powder without labeling and they will not be aware of which they receive (egg white or whole egg).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole egg powder (Experimental): Participants are given whole egg powder which contains high levels of the nutrients choline, lutein, and docosahexaenoic acid.
  Interventions: Dietary Supplement: Whole Egg Powder
- Egg white powder (Placebo Comparator): The participants are given an egg white powder that does not contain the target nutrients (choline, lutein, and docosahexaenoic acid).
  Interventions: Dietary Supplement: Egg White Powder

INTERVENTIONS:
Dietary Supplement: Whole Egg Powder — Breastfeeding mothers will consume the equivalent of 5 whole eggs per week for 3 months.
  Arms: Whole egg powder
Dietary Supplement: Egg White Powder — Breastfeeding mothers will consume the equivalent of 5 egg whites per week for 3 months.
  Arms: Egg white powder

SUMMARY:
Purpose: To establish a whole food, egg, as a viable study material to supplement mothers and infants with nutrients that support optimal brain development. There will be 84 breastfeeding dyads, 3 months postnatal.

Mothers will be randomized to a whole egg or egg white (due to lack of an appropriate control food). Initial diet intake will be screened using the NDSR. Participants will come to the lab 3 times across 3 months (age 3 months, 4.5 months, and 6 months). Milk, saliva, and plasma will be collected from the mother, while saliva and plasma (heel stick) are collected from the infant. Diet data will be collected at each visit. The infant will complete a recognition memory test using electrophysiology at 6 months as well as the Bayley Scales of Infant Development at 4.5 months. The mother will complete a temperament questionnaire at 3 months and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* infant is 12-15 weeks of age at enrollment
* healthy, lactating mother age 18-35
* gave birth at >38 weeks gestation without remarkable incident
* consuming <=50% of the recommended amounts of 2 of the 3, DHA, choline, and lutein

Exclusion Criteria:

* infant with diagnosis or documented suspicion of developmental delay
* egg allergy or family history of egg allergy
* gestational diabetes
* any documented seizure activity

Ages: 3 Months to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 84 (Estimated)
Dates: Start 2019-02-05 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Recognition Memory in an Oddball Task | 13 weeks (at 6 months of age)
  The difference in microvolts between the negative deflection to novel pictures and the negative deflection to familiar pictures at approximately 100-400ms after the pictures come on the screen will be measured in an event-related potentials (ERP) paradigm. The investigators hypothesize that the whole egg group will have better memory for the familiar pictures than the egg white group.

OTHER OUTCOMES:
Bayley Scales of Infant Development (BSID) | 6 weeks (at 4.5 months of age)
  BSID administered at 4.5 months

CONTACTS AND LOCATIONS:
Overall Officials: Carol L Cheatham, Ph.D., Principal Investigator — Associate Professor, University of North Carolina-Chapel Hill
Locations (1):
- Nutrition Research Institute, Kannapolis, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No